CLINICAL TRIAL: NCT06651879
Title: The Preoperative Use of Ultrasound in Airway Assessment in Critically Ill Obstetrics with Pre-eclampsia; Comparison Between Two Ultrasound Techniques in Relation to the Standard Clinical Assessment
Brief Title: Ultrasound Airway Assessment of Critically Ill Preeclamptic; Comparison Between Two Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FMASU R147/2024
Record Dates: First submitted 2024-08-02; First posted 2024-10-22 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Critical Illness; Difficult; Intubation, Postpartum, During Puerperium; Pre-Eclampsia
MeSH Terms: conditions — Critical Illness; Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: The trial is a pilot of randomized clinical, two parallel groups, 1:1 allocation, superiority study.
Who Masked: Care Provider
Masking Description: both care providers are blinded: the ultrasound examiner will be blinded regarding the clinical evaluation of the airway.
  the anesthesiologist will be blinded regarding the ultrasound airway assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two views ultrasound technique (Experimental): : the ultrasound examiner will use the difficult airway examination by sonography (DARES) protocol in which involves only two views of the upper airway: the thyrohyoid and the suprahyoid views. Measurements selected for this protocol include the DSE, HMD, HMDR1, HMDR2, and tongue thickness, which cover all three domains of TTD, APD, and OSD
  Interventions: Diagnostic Test: techniques of ultrasound examination of the airway
- Five views ultrasound technique (Active Comparator): The thicknesses of the anterior neck soft tissues will be measured by systematic examination includes five views: 1) Suprahyoid View .2) Thyrohyoid view; will be used to visualize epiglottis and pre -epiglottic space(PES).3) Thyroid view; for vocal cord visualization.4) Cricothyroid view .5) Suprasternal view From the previous views the following will be measured: tongue volume (TV ) ANS-H: anterior neck skin thickness at hyoid; TMD: thyromental distance; ANS-E: anterior neck skin thickness at epiglottis; ANS-VC: anterior neck skin thickness at vocal cords; SD: subglottic diameter PreE: pre epiglottic space; aVF: anterior vocal folds; pVF: posterior vocal folds; mVF: midpoint of anterior , posterior vocal folds , and diameter of the transverse tracheal air shadow in the subglottic area . The following will be calculated PreE/aVF, PreE/mVF , PreE/pVF and PreE/E-VC. That will be in addition to detection of any abnormalities in the airway
  Interventions: Diagnostic Test: techniques of ultrasound examination of the airway

INTERVENTIONS:
Diagnostic Test: techniques of ultrasound examination of the airway — two different techniques of ultrasound. The techniques are the two views and the five views

SUMMARY:
Unexpected difficult airway exposes the patient to serious morbidity and even mortality. The changes in pregnancy and preeclampsia increase the risk of difficult intubation. Proper anticipation affects the outcome and enhances safety, especially in critically ill patients. This research aims to assess the superiority of either 2 views or 5 views ultrasound assessment in predictivity of difficult airway (difficult ventilation, laryngoscopy, and intubation) and their comparison to traditional clinical examination by El-Ganzouri Risk Index (EGRI) in critically ill obstetric patients with pre-eclampsia.

DETAILED DESCRIPTION:
Unexpected difficult airway exposes the patient to serious morbidity and even mortality. Obstetrics airway carries the risk of complications due to physiological changes. The airway shows more restriction and changes in preeclamptic patients and peripartum periods. A study reported one incidence of difficult intubation in obstetrics in 20 cases. Inadequate airway management leads to failure in ventilation and oxygenation of the critically ill mother and her fetus.

the Practice Guidelines for Management of the Difficult Airway by the American Society of Anesthesiologists (ASA) define the difficult airway as difficult facemask ventilation of the upper airway, difficult tracheal intubation, or both. preoperative assessment of the airway avoids that risk; however, current clinical screening tests have low sensitivity and specificity with limited predictivity.

Ultrasound (US) provides a more precise assessment for tissues like epiglottis, vocal cords, and ring-shaped membranes; thus, it facilitates a bedside, non-invasive objective airway assessment. Moreover, ultrasound assessment can plan and guide airway interventions if needed. The airway in pregnancy goes through changes. a study concluded that The US airway assessment parameters differ significantly between pregnant and non-pregnant patients. Previous studies reported that the best predictors of difficult laryngoscopy and/or difficult intubation were the epiglottis midline-skin distance, hyoid bone-to-skin distance, thyroid cartilage-to-skin distance, thyrohyoid membrane-to-skin distance, and vocal cord anterior commissure-skin distance also predicted difficult airway. In Pregnancy, hyoid bone visibility, and Pre-E/E-VC ratio were independent predictors of the difficult airway.

Researchers suggested different techniques for airway ultrasound. Some suggested detailed technique that allows the determination of multiple parameters. Others suggested a more concise protocol to lessen the time of assessment and to avoid complexity.

This trial assesses the superiority of either 2 views or 5 views ultrasound assessment in predictivity of difficult airway (difficult ventilation, laryngoscopy, and intubation) and their comparison to traditional clinical examination by El-Ganzouri index (GREI) (9) in critically ill obstetric patients with pre-eclampsia.

ELIGIBILITY:
Inclusion Criteria:Critically ill preeclamptic patients for caesarean section under general anesthesia with the following criteria:

* Aged from 18 to 60 years.
* Singleton or multiple pregnancies,
* Mentally competent.
* American Society of Anesthesiologists (ASA) physical status I, II and III

Exclusion Criteria:

* Patient's Refusal to participate,
* Abnormal pharynx or airway anatomy,
* expected difficult laryngoscopy with cervical spine abnormality,
* Maxillofacial anomalies,
* upper airway diseases or malignancy,
* Unconscious women,
* those with learning difficulties, or mentally handicapped

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-20 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
The predictivity of both us techniques in relation to clinical assessment of El-Ganzouri index (EGRI). | the degree of difficult intubation will be assesed intraoperative after aneesthesia and intubation, clinical assessment will be preoperative, the us assessment will be preoperative at the same day of operation or immediately postoperative
  Sensitivity and specificity of the measured parameters in both ultrasound techniques in relation to the clinical El-ganzouri score where (score < 4 is unlikely to be difficult and score ≥ 4 is more likely to be difficult) to predict difficult airway.
The predictive superiority between 2 view and 5 views ultrasound techniques regarding difficult ventilation, laryngoscopy and intubation | the actual degree of difficult intubation will be assesed intraoperative after aneesthesia and intubation, the us assessment will be done preoperative at the same day of operation or immediately postoperative
  * Difficult ventilation is measured by Hans score where grade 0 and 1 will be categorized as easy ventilation, while <= 2 are difficult
  * Difficult intubation is measured by Cormack-Lehane grade where where grade 1 nad 2a will be categorized as easy while <= 2b will be categorized as difficult.
  * Prolonged intubation <10 min or repeated attempts < 3 will be categorized as difficult.

SECONDARY OUTCOMES:
postoperative side effects | within 24 hours postoperative
  Any postoperative adverse effects as patient discomfort from airway, mandibular pain or stridor
duration of the airway assessment | preoperative
  time needed for ultrasound evaluation measured from the start of the technique till the end of the ultrasound examination, and duration of the clinical EL-Ganzouri assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gomes SH, Simoes AM, Nunes AM, Pereira MV, Teoh WH, Costa PS, Kristensen MS, Teixeira PM, Pego JM. Useful Ultrasonographic Parameters to Predict Difficult Laryngoscopy and Difficult Tracheal Intubation-A Systematic Review and Meta-Analysis. Front Med (Lausanne). 2021 May 28;8:671658. doi: 10.3389/fmed.2021.671658. eCollection 2021. PMID 34124099
- [Background] Zheng BX, Zheng H, Lin XM. Ultrasound for predicting difficult airway in obstetric anesthesia: Protocol and methods for a prospective observational clinical study. Medicine (Baltimore). 2019 Nov;98(46):e17846. doi: 10.1097/MD.0000000000017846. PMID 31725624
- [Background] Izci B, Riha RL, Martin SE, Vennelle M, Liston WA, Dundas KC, Calder AA, Douglas NJ. The upper airway in pregnancy and pre-eclampsia. Am J Respir Crit Care Med. 2003 Jan 15;167(2):137-40. doi: 10.1164/rccm.200206-590OC. Epub 2002 Oct 31. PMID 12411285
- [Background] Bala R, Budhwar D, Kumar V, Singhal S, Kaushik P, Sharma J. Clinical and ultrasonographic assessment of airway indices among non-pregnant, normotensive pregnant and pre-eclamptic patients: a prospective observational study. Int J Obstet Anesth. 2023 May;54:103637. doi: 10.1016/j.ijoa.2023.103637. Epub 2023 Feb 1. PMID 36827944